CLINICAL TRIAL: NCT00953862
Title: Efficacy of Atomoxetine in Adults With ADHD and Substance Abuse Disorder Being Treated in a Residential Treatment Facility
Brief Title: Atomoxetine/Attention Deficit/ Hyperactive Disorder (ADHD)/Substance Use Disorder (SUD)in a Residential Treatment Facility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#12233; BAZ-US-X031
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Substance Use Disorder; Residential Treatment Facility
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Substance-Related Disorders | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atomoxetine Treatment Arm (Experimental): Patients who were identified as having adult ADHD on the ACDS were offered an open label treatment trial with atomoxetine, up to 120 mg/day over 10 weeks. Atomoxetine was titrated over a period of four weeks based upon clinical response and observed side-effects. All patients receiving atomoxetine gave written informed consent prior to participation and were assessed for ADHD symptoms via the Adult Investigator Adult ADHD Symptom Rating Scale (AISRS) every 1-2 weeks. All patients received a physical exam, review of systems and routine blood work prior to treatment. Data were analyzed for patients completing at least 2 weeks of atomoxetine therapy. Treatment response was pre-hoc defined as having a >=30% reduction in total AISRS scores from baseline.
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — In Phase II, atomoxetine was dispensed beginning at 25 mg/day. Dose was adjusted based on clinical response and tolerability over a 4-week period up to 120mg/day and held constant at the optimized level for the final 6 weeks of the trial.

SUMMARY:
Although Attention Deficit/ Hyperactive Disorder (ADHD) is a common comorbidity in individuals diagnosed with Substance Use Disorder (SUD), little data currently exists on the utility of screening tools in large samples of adult patients with SUD in inpatient treatment. This was a 10-week, 2-phase, open label trial of atomoxetine for ADHD in adult patients being treated for a co-morbid SUD in a residential treatment facility (RTF). The primary objective of the study was to assess the efficacy of atomoxetine in adults with an SUD and ADHD. Secondary objects included assessment of the co-morbidity of ADHD and the safety and tolerability of atomoxetine in this population.

DETAILED DESCRIPTION:
Phase 1: Patients with SUD who were either newly admitted (abstinent for <1 week) or in treatment in the RTF (abstinent <3 months) were administered the Adult ADHD Self-Report Scale Symptom Checklist (ASRS) v. 1.1 Screener. Patients who screened positive(>= 4 out 6 significant items) were then administered the Adult Clinician Diagnostic Scale (ACDS) v.1.2 to establish a diagnosis of ADHD and the Predictive Value Positive (PVP) in this population.

Phase II (Treatment): Participants who screened positive for ADHD on the ACDS were given informed consent and baseline evaluations for inclusion. Those meeting inclusion/exclusion criteria were treated with atomoxetine starting at 25 mg/day. The dose was adjusted based on clinical response and tolerability over a 4-week period up to 120 mg/day and held constant for the final six weeks of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Are between the ages of 18-60, inclusive.
2. Meet diagnostic criteria for substance dependence.
3. Meet Diagnostic and Statistics Manual of Mental Disorders-IV (DSM-IV) criteria for attention deficit hyperactivity disorder as assessed by the Adult ADHD Clinician Diagnostic Scale (ACDS).
4. Must be able to communicate effectively with the investigator and study staff.
5. Must be able to swallow capsules.
6. Reside at Odyssey House for duration of study.

Exclusion Criteria:

1. Lifetime or present history of bipolar disorder, schizophrenia or schizoaffective disorder. Assessment will be made by comprehensive psychiatric diagnostic interview.
2. Have organic brain disease (such as dementia) or traumatic brain injury residua. Have a history of seizure disorder (other than febrile seizures) or patients who have taken (or are currently taking) anticonvulsants for seizure control.
3. Females who are currently pregnant or breast feeding, and women of child-bearing potential who are not currently using an adequate form of birth control.
4. Medical conditions limiting participation in the study.
5. Patients who are at serious suicidal or homicidal risk.
6. Have significant prior or current medical conditions that could be exacerbated or compromised by atomoxetine.
7. Who have glaucoma.
8. Have a history of difficulty starting a stream of urine or other symptoms suggestive of prostate enlargement.
9. Who anticipate moving or traveling extensively during the study period.
10. Have a medical condition that would, in the opinion of the study physician, make participation medically hazardous.
11. Be anyone who in the opinion of the investigator would not be expected to complete the study protocol due to probable incarceration or relocation from the clinic area.

    -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2005-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lenard Adler, MD, Principal Investigator — NYU School of Medicine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were adult Odyssey House residents who met DSM-IV criteria for ADHD based on the Adult ADHD Clinician Diagnostic Scale v1.2 (ACDS v1.2) and drug and/or alcohol dependence based on Structured Clinical Interview for DSM Disorders - Patient Edition (SCID-I/P). Study was conducted from July 2005 to February 2007.
Pre-assignment Details: Patients were excluded if they had a diagnosis of bipolar disorder, schizophrenia or schizoaffective disorder, as assessed by clinical history and the SCID-I/P; seizure history (other than febrile seizures); current chronic or acute illness or medical condition, glaucoma, organic brain disease, traumatic brain injury, pregnancy, or lactation.
Groups:
- Atomoxetine Arm: Patients who were identified as having adult ADHD on the ACDS were offered an open label treatment trial with atomoxetine, up to 100 mg/day over 10 weeks. Atomoxetine was titrated over a period of four weeks based upon clinical response and observed side effects. All patients receiving atomoxetine gave written informed consent prior to participation and were assessed for ADHD symptoms via the Adult Investigator Adult ADHD Symptom Rating Scale (AISRS) every 1-2 weeks. All patients received a physical exam, review of systems and routine blood work prior to treatment. Data were analyzed for patients completing at least 2 weeks of atomoxetine therapy. Treatment response was pre-hoc defined as having a >=30% reduction in total AISRS scores from baseline.
  Atomoxetine : In Phase II, atomoxetine was dispensed beginning at 25 mg/day. Dose was adjusted based on clinical response and tolerability over a 4-week period up to 120mg/day and held constant for the final 6 weeks of the trial.
Period: Overall Study
Arm/Group | Atomoxetine Arm
Started | 18
Completed | 12
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: This number is the total number who were found eligible for the treatment.
Groups:
- Treatment: Patients who were identified as having adult ADHD on the ACDS were offered an open label treatment trial with atomoxetine, up to 100 mg/day over 10 weeks. Atomoxetine was titrated over a period of four weeks based upon clinical response and observed side effects. All patients receiving atomoxetine gave written informed consent prior to participation and were assessed for ADHD symptoms via the Adult Investigator Adult ADHD Symptom Rating Scale (AISRS) every 1-2 weeks. All patients received a physical exam, review of systems and routine blood work prior to treatment. Data were analyzed for patients completing at least 2 weeks of atomoxetine therapy. Treatment response was pre-hoc defined as having a >=30% reduction in total AISRS scores from baseline.
  Atomoxetine : In Phase II, atomoxetine was dispensed beginning at 25 mg/day. Dose was adjusted based on clinical response and tolerability over a 4-week period up to 120mg/day and held constant for the final 6 weeks of the trial.
Arm/Group | Treatment
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  African-American | 12
  Caucasian | 3
  Hispanic | 3
Substance Used [Number; unit: Participants]
  Cocaine | 6
  Cannabis | 5
  Alcohol | 3
  Opioid | 3
  Other/Unable to report | 1
Length of Abstinence from all Substances [Mean (Standard Deviation); unit: Weeks] | 14.1 (18.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Adult ADHD Investigator Symptom Rating Scale Score
Description: The AISRS (Adult ADHD Investigator Symptom Rating Scale) consists 18-items that directly correspond to the 18 DSM-IV symptoms of ADHD. Each item is scored on a 4-point scale (0 = none; 1 = mild; 2 = moderate; and 3 = severe, higher score is more impaired). The total summed score was at minimum 0 and at maximum 54 (the higher the score the more severe the symptomatology).
Time Frame: Baseline and week 10 of treatment
Population: Those treated with atomoxetine who were not discontinued due to receiving less than 2 weeks of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine Arm
Number analyzed (Participants) | 12
units on a scale | 17.3 (11.9)

2. Secondary Outcome: Change in Adult ADHD Symptom Rating Scale v1.1 Symptom Checklist Score
Description: The ASRS (Adult ADHD Symptom Rating Scale) v1.1 Symptom Checklist is an 18-item scale developed by the workgroup on Adult ADHD for the World Health Organization designed to assess the frequency of ADHD symptoms on a 0-4 scale (0 = never, 1 = rarely, 2 = sometimes, 3= often, and 4 = very often, minimum total summed score of 0 and maximum total summed score of 72, higher score is more impairment).
Time Frame: Baseline and week 10 of treatment
Population: Those treated with atomoxetine who were not discontinued due to receiving less than 2 weeks of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Atomoxetine Phase: Patients who were identified as having adult ADHD on the ACDS were offered an open label treatment trial with atomoxetine, up to 100 mg/day over 10 weeks. Atomoxetine was titrated over a period of four weeks based upon clinical response and observed side effects. All patients receiving atomoxetine gave written informed consent prior to participation and were assessed for ADHD symptoms via the Adult Investigator Adult ADHD Symptom Rating Scale (AISRS) every 1-2 weeks. All patients received a physical exam, review of systems and routine blood work prior to treatment. Data were analyzed for patients completing at least 2 weeks of atomoxetine therapy. Treatment response was pre-hoc defined as having a >=30% reduction in total AISRS scores from baseline.
  Atomoxetine : In Phase II, atomoxetine was dispensed beginning at 25 mg/day. Dose was adjusted based on clinical response and tolerability over a 4-week period up to 120mg/day and held constant for the final 6 weeks of the trial.
Arm/Group | Atomoxetine Phase
Number analyzed (Participants) | 12
units on a scale | 19.7 (18.7)

3. Secondary Outcome: Change in Clinical Global Impression-- Severity of Illness Score
Description: The CGI-S (Clinical Global Impression-- Severity of Illness) scale is a single-item rating scale of the clinician's assessment of the global severity of ADHD symptoms in relation to the clinician's total experience with ADHD patients. Severity is rated on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill).
Time Frame: Baseline and week 10 of treatment
Population: Those treated with atomoxetine who were not discontinued due to receiving less than 2 weeks of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine Arm
Number analyzed (Participants) | 12
units on a scale | 1.1 (0.9)

ADVERSE EVENTS:
Description: The study results analyses for adverse events did not specify what "other" meant and will therefore be only presented as "other" without specification.
Groups:
- Treatment Phase: Patients who were identified as having adult ADHD on the ACDS were offered an open label treatment trial with atomoxetine, up to 100 mg/day over 10 weeks. Atomoxetine was titrated over a period of four weeks based upon clinical response and observed side effects. All patients receiving atomoxetine gave written informed consent prior to participation and were assessed for ADHD symptoms via the Adult Investigator Adult ADHD Symptom Rating Scale (AISRS) every 1-2 weeks. All patients received a physical exam, review of systems and routine blood work prior to treatment. Data were analyzed for patients completing at least 2 weeks of atomoxetine therapy. Treatment response was pre-hoc defined as having a >=30% reduction in total AISRS scores from baseline.
  Atomoxetine : In Phase II, atomoxetine was dispensed beginning at 25 mg/day. Dose was adjusted based on clinical response and tolerability over a 4-week period up to 120mg/day and held constant for the final 6 weeks of the trial.
Arm/Group | Treatment Phase
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 9/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase (N=18)
Headache (Vascular disorders) | 2
Abdominal pain/cramps (Gastrointestinal disorders) | 2
Other (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No